CLINICAL TRIAL: NCT00665353
Title: A Pilot Study of Therapy With Pioglitazone Prior to HCV Treatment in HIV-1 and HCV Genotype 1-Infected Subjects With Insulin Resistance Who Are Prior Nonresponders to Peginterferon and Ribavirin Therapy
Brief Title: Pioglitazone Before Peginterferon and Ribavirin for Hepatitis C Infection in HIV/HCV-Coinfected Patients With Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5239; 1U01AI068636 (NIH); NCT00735982 (obsolete NCT alias)
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV-1 and Hepatitis C Co-Infection
Keywords: HIV; HCV
MeSH Terms: interventions — Pioglitazone; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PIO (step 1) then PIO+PEG-INF+RBV (step 2) (Experimental): All participants in this study will receive pioglitazone therapy for 24 to 28 weeks. Participants will continue pioglitazone and add peginterferon and ribavirin to their treatment regimen for up to 48 additional weeks.
  Interventions: Drug: pioglitazone; Drug: peginterferon; Drug: ribavirin

INTERVENTIONS:
Drug: pioglitazone — Traditionally used in the treatment of type 2 diabetes to increase insulin sensitivity. Participants will take 30 mg daily in tablet form.
Drug: peginterferon — Used in the treatment of HCV. Participants will receive 180 mcg subcutaneously once a week.
Drug: ribavirin — Used in the treatment of HCV. Participants will receive 1000 to 1200 mg orally per day depending on weight.

SUMMARY:
Insulin resistance is common in people coinfected with HIV and Hepatitis C virus (HCV) and is associated with poor responses to treatment for HCV. Pioglitazone is an FDA-approved medication for the treatment of type 2 diabetes. It works by increasing the body's sensitivity to insulin. The purpose of this study is to determine whether treatment with pioglitazone prior to HCV treatment with peginterferon and ribavirin is safe and effective in improving the treatment outcome in insulin-resistant, HIV/HCV-coinfected people for whom previous treatment with peginterferon and ribavirin was unsuccessful.

DETAILED DESCRIPTION:
New and better strategies for the treatment of HCV in HIV/HCV-coinfected people are urgently needed. Standard therapy for HCV includes treatment with peginterferon plus ribavirin. Peginterferon is a modified form of the drug interferon and is used either alone or in combination with ribavirin for the treatment of HCV. Ribavirin works by stopping HCV from multiplying inside the body. Sustained virologic response rates in past large studies of peginterferon plus ribavirin used for treating HCV types 1 or 4 ranged from 11% to 29%. Studies have shown that insulin resistance in HCV-infected people who are HIV uninfected leads to poorer HCV treatment response. Improving the body's response to insulin may also improve the outcome of treatment for HCV.

Participants in this study will take pioglitazone alone for up to 28 weeks. At Entry and Weeks 2, 4, 8, 12,18, and 24 participants will receive clinical assessments. At Week 24, participants will undergo additional tests to ensure that they can enter Step 2 of the study. Participants who are able to continue will then take peginterferon and ribavirin in addition to the pioglitazone for up to 48 additional weeks. Clinical assessments will take place at the time of entry and Weeks 2, 4, 8, 12, 16, and 24 of Step 2. Participants who do not exhibit a response to the treatment at Weeks 12 or 24 will not continue Step 2, as it is unlikely that further treatment will elicit a response. Participants who continue in the study will return to the study site for clinical assessments at Weeks 32, 40, and 48 of Step 2. Follow-up visits will be held at Weeks 60 and 72. The assessments done at clinic visits may include any or all of the following tests: thyroid function, hematology and chemistry, fasting plasma glucose, liver function, gamma-glutamyl transferase, pregnancy, CD4/CD8, HIV-1 RNA, qualitative HCV RNA, and quantitative HCV RNA.

On November 18, 2011 the study was closed to accrual due to not meeting targeted accrual goals.

ELIGIBILITY:
Inclusion Criteria:

For Step 1:

* HIV infected
* Exhibited no response to previous treatment with PEG-IFN alfa-2a 180 mcg/week or alfa-2b 1.5 mcg/kg/week and at least 1000 mg/day ribavirin given for at least 12 consecutive weeks. More information on this criterion can be found in the protocol.
* HOMA-IR valued greater than 2.5 within 42 days prior to study entry. More information on this criterion can be found in the protocol.
* CD4 count of at least 200 cells/mm3 within 42 days prior to study entry
* HCV RNA of at least 60 IU/ml by quantitative RT-PCR assay with or without reactive anti-HCV antibodies within 42 days prior to study entry
* Documentation of infection with HCV genotype 1, within 42 days prior to study entry
* On stable or no antiretroviral therapy for 12 weeks prior to study entry. Interruptions in treatment lasting 14 days or less are allowed if the participant reinitiated the same regimen prior to study entry. Dose modifications or changes in drug formulations during the 12 weeks prior to study entry are permissible.
* Participants on antiretroviral therapy should plan to remain on the same therapy for at least 24 weeks after study entry. Participants not on antiretroviral therapy should have no plans to initiate therapy during the first 24 weeks following study entry.
* Participants with documented or suspected hepatic cirrhosis must have a modified Child-Pugh-Turcotte (CPT) within 42 days prior to study entry.
* Participants with documented or suspected hepatic cirrhosis must have either serum alpha-fetoprotein level of 50 ng/ml or less within 24 weeks prior to study entry; OR serum alpha-fetoprotein greater than 50 ng/ml but no greater than 400 ng/ml with an imaging procedure that shows no evidence of a hepatic tumor, both obtained within 24 weeks prior to study entry.
* Certain laboratory values obtained within 42 days prior to study entry. More information on this criterion can be found in the protocol.
* Willing to use effective forms of contraception throughout the study. More information on this criterion can be found in the protocol.
* Ability and willingness of participant to give written informed consent.

For Step 2:

* No more than 28 days have passed since the Step 1, Week 24 visit
* Participants who were treated in Step 1 who meet the following criteria:

  1. Detectable HCV RNA (> 60 IU/mL) at the Step 1, Week 24 evaluation
  2. CD4 cell count of at least 200 cells/mm3 at Week 24. If the CD4 count is less than 200 cells/mm3 at Week 24, then it must not have decreased by more than 20 cells/mm3 from the Step 1 entry value.
  3. Taking pioglitazone at the time of Step 2 entry
* Certain laboratory values obtained within 28 days prior to Step 2 entry. More information on this criterion can be found in the protocol.
* Willing to use an effective form of contraception throughout the study
* Female participants of reproductive potential are required to have a negative serum or urine β-HCG pregnancy test within 14 days prior to Step 2 entry
* Participants without a pregnant partner.

Exclusion Criteria:

* Presence of known causes of significant liver disease. More information on this criterion can be found in the protocol.
* Evidence of decompensated liver disease manifested by presence or history of ascites, variceal bleeding, or hepatic encephalopathy
* History of HCV treatment within 28 days prior to study entry
* Evidence that nonresponse to prior HCV treatment may have been due to nonadherence or certain dose reductions. More information on this criterion can be found in the protocol.
* Use of interferon gamma, TNF-alpha inhibitors, rifampin, rifabutin, pyrazinamide, isoniazid, ganciclovir, or hydroxyurea within 14 days prior to study entry
* Current use of didanosine or zidovudine or plans to initiate use of either during the study
* Active drug or alcohol abuse or dependence that, in the opinion of the study investigator, could interfere with adherence to study requirements
* History of uncontrolled seizure disorder
* Uncontrolled depression or other psychiatric disorder, such as untreated Grade 3 psychiatric disorder, Grade 3 disorder not amenable to medical intervention, or any hospitalization within the past 52 weeks that may affect tolerability of study requirements
* History of autoimmune disorders, including but not limited to Crohn's disease, ulcerative colitis, severe psoriasis, and rheumatoid arthritis, that have been exacerbated by previous interferon use
* Any systematic antineoplastic or immunomodulatory treatment or radiation within 24 weeks prior to study entry
* Serious illness including malignancy, active symptomatic coronary artery disease within 24 weeks prior to study entry, or other chronic medical condition that could interfere with safe study completion
* Presence of AIDS-defining opportunistic infections within 12 weeks prior to study entry
* Hemoglobinopathy (e.g., thalassemia major) or any other cause of or tendency to hemolysis. Subjects with thalassemia minor may be enrolled at the discretion of the investigator.
* History of major organ transplantation with an existing functional graft
* Use of antidiabetic medications for any reason within 12 weeks prior to study entry
* Fasting plasma glucose level of at least 126 mg/dl within 42 days prior to study entry or current or previous treatment at any time for diabetes with measures other than diet. Women with a history of gestational diabetes, patients with diabetes or hyperglycemia occurring in the context of short term use of corticosteroids, growth hormone, or other diabetogenic medication, and patients with diabetes or hyperglycemia following an episode of pancreatitis who no longer require treatment for diabetes are not excluded.
* Known osteoporosis or receipt of treatment of osteopenia or osteoporosis within 12 weeks prior to study entry with the following medications: risedronate (Actonel®), ibandronate (Boniva®), etidronate (Didronel®), raloxifene (Evista®), teriparatide (Forteo®), aledronate (Fosamax®), calcitonin (Miacalcin®).
* Known initiation or change in dose of any statins, fibrates, omega-3 fatty acids, bile acid sequestrants, ezetimibe, and niacin derivatives within 12 weeks prior to study entry
* Known allergy, sensitivity, or hypersensitivity to components of the study drugs or their formulation
* Regular and excessive use of alcohol within the 12 weeks prior to study entry. More information on this criterion can be found in the protocol.
* Unwilling to restrict alcohol use during the study to 120 g of alcohol per week or less for men and 60 g of alcohol per week or less for women
* Known glucocorticoid use in supraphysiologic doses (e.g., more than 10 mg per day of prednisone or equivalent doses of other glucocorticoids) within 12 weeks prior to study entry
* Known glucocorticoid use in physiologic replacement doses (e.g., 10 mg or less per day of prednisone or equivalent doses of other glucocorticoids) initiated within 28 days prior to study entry
* History of congestive heart failure corresponding to New York Heart Association Class II or greater
* Current use of prohibited concomitant medications. More information on this criterion is available in the protocol.
* Current participation in experimental studies that include treatments not approved by the FDA or any blinded treatments, with the exception of investigational antiretrovirals available through expanded access programs
* Body mass index (BMI) greater than 35 kg/m2
* Participant or participant's partner is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Glesby, MD, PhD, Study Chair — Cornell Clinical Trials Unit, Weill Medical College of Cornell University; Kristen Marks, MD, MS, Principal Investigator — New York Presbyterian Hospital-Cornell
Locations (8):
- United States (8):
  - Ucsf Aids Crs (801), San Francisco, California
  - Northwestern University CRS (2701), Chicago, Illinois
  - New Jersey Medical School-Adult Clinical Research Ctr. CRS (31477), Newark, New Jersey
  - Cornell CRS (7804), New York, New York
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - AIDS Care CRS (1108), Rochester, New York
  - Metro Health CRS (2503), Cleveland, Ohio
  - Virginia Commonwealth Univ. Medical Ctr. CRS (31475), Richmond, Virginia

REFERENCES:
- [Background] de Larranaga GF, Wingeyer SD, Puga LM, Alonso BS, Benetucci JA. Relationship between hepatitis C virus (HCV) and insulin resistance, endothelial perturbation, and platelet activation in HIV-HCV-coinfected patients under highly active antiretroviral treatment. Eur J Clin Microbiol Infect Dis. 2006 Feb;25(2):98-103. doi: 10.1007/s10096-006-0090-6. PMID 16477441
- [Background] Patel MR, Mullen MP, Dieterich DT. Sustained virologic response with short-course ribavirin and peginterferon treatment in 2 patients coinfected with HIV and HCV genotype 1. AIDS Read. 2006 Mar;16(3):164, 168-9; discussion 168-9. PMID 16538956
- [Background] Romero-Gomez M, Del Mar Viloria M, Andrade RJ, Salmeron J, Diago M, Fernandez-Rodriguez CM, Corpas R, Cruz M, Grande L, Vazquez L, Munoz-De-Rueda P, Lopez-Serrano P, Gila A, Gutierrez ML, Perez C, Ruiz-Extremera A, Suarez E, Castillo J. Insulin resistance impairs sustained response rate to peginterferon plus ribavirin in chronic hepatitis C patients. Gastroenterology. 2005 Mar;128(3):636-41. doi: 10.1053/j.gastro.2004.12.049. PMID 15765399
- [Background] Torriani FJ, Rodriguez-Torres M, Rockstroh JK, Lissen E, Gonzalez-Garcia J, Lazzarin A, Carosi G, Sasadeusz J, Katlama C, Montaner J, Sette H Jr, Passe S, De Pamphilis J, Duff F, Schrenk UM, Dieterich DT; APRICOT Study Group. Peginterferon Alfa-2a plus ribavirin for chronic hepatitis C virus infection in HIV-infected patients. N Engl J Med. 2004 Jul 29;351(5):438-50. doi: 10.1056/NEJMoa040842. PMID 15282351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 8 ACTG sites. The dates of first and last study enrollments were March 31, 2009 and May 26, 2010, respectively.
Pre-assignment Details: A5239 was a single-arm study which enrolled prior nonresponders to peginterferon (PEG-IFN) and ribavirin (RBV)> therapy with documented insulin resistance. 31 potential subjects failed to meet all inclusion/exclusion criteria. 22 of these potential subjects did not meet the HOMA-IR criterion (> 2.5 within 42 days prior to study entry).
Groups:
- PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2): All participants in Step 1 received pioglitazone therapy for 24 to 28 weeks. Participants continued pioglitazone and add peginterferon and ribavirin to their treatment regimen for up to 48 additional weeks in Step 2.
Period: Study Step 1
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Started | 19
Completed | 16
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Period: Study Step 2
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Started | 16
Completed | 2
Not Completed | 14
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 12

BASELINE CHARACTERISTICS:
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants] — Derived from self-reported race and ethnicity.
  participants
    White non-Hispanic | 8
    Black non-Hispanic | 9
    Hispanic (regardless of race) | 2
Region of Enrollment [Number; unit: participants]
  United States | 19
Age categorical [Number; unit: participants]
  30 - 39 years | 1
  40 - 49 years | 9
  50 - 59 years | 8
  60 - 69 years | 1
IV drug history [Number; unit: participants] — Self-reported
  participants
    Never | 7
    Previously | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (weight in kilograms divided by height in meters squared)
  kg/m^2 | 27.7 (4.1)
HIV-1 RNA [Number; unit: participants]
  < 50 copies/mL | 15
  50 - 99 copies/mL | 2
  100 - 499 copies/mL | 2
CD4 count [Mean (Standard Deviation); unit: cells/mm^3] | 567 (192)
Nadir CD4 count [Number; unit: participants]
  <= 50 cells/mm^3 | 4
  51 - 100 cells/mm^3 | 4
  101 - 200 cells/mm^3 | 4
  201 - 500 cells/mm^3 | 6
  > 500 cells/mm^3 | 1
Thyrotropin [Mean (Standard Deviation); unit: mIU/L] — N=17, 2 were missing results
  mIU/L | 1.49 (0.67)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.4 (1.5)
Absolute neutrophil count [Mean (Standard Deviation); unit: cells/mm^3] | 2501 (1031)
Platelets [Mean (Standard Deviation); unit: cells/mm^3] | 185842 (67375)
Direct bilirubin [Mean (Standard Deviation); unit: * ULN] | 1.0 (0.6)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: * ULN] | 1.4 (1.2)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: * ULN] | 1.5 (0.9)
Gamma-glutamyl transferase [Mean (Standard Deviation); unit: U/L] — N=14, 5 had missing results.
  U/L | 154 (127)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 100 (12)
Fasting insulin [Mean (Standard Deviation); unit: mIU/L] | 25 (13)
Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: mg/dL x mIU/L / 405] | 6.3 (3.5)
Prior hepatitis C virus (HCV) non-response type [Number; unit: participants]
  < 2 log10 drop AND detectable >= 10 and < 22 weeks | 13
  Detectable after >= 22 and < 30 weeks | 6

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of All Subjects With HCV Viral Load < 60 IU/mL at Week 24 of Step 2.
Time Frame: Week 24 of Step 2
Population: All enrolled subjects.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 19
proportion of participants | 0.158 [0.059 to 1]
Statistical Analysis 1: Comparison: PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2); The proportion of subjects responding was compared to a historical null rate of 0.10. The hypothesized response rate was 0.30; Test type: Superiority or Other; p = 0.29, Exact test of proportions — This is an unadjusted p-value. Statistical significance was defined a priori as 0.10; proportion = 0.158, 90% CI 1-sided [lower limit 0.059]

2. Secondary Outcome: Safety and Tolerability
Description: Summary of the number of subjects with at least one grade 3 or higher sign/symptom or laboratory abnormality.
Time Frame: Step 1 (Up to 24 to 28 weeks)
Population: All enrolled subjects.
Measure: Number; unit: participants
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 19
participants | 7

3. Secondary Outcome: Safety and Tolerability
Description: Summary of the number of subjects with at least one grade 3 or higher sign/symptom or laboratory abnormality.
Time Frame: Step 2 (Up to 72 weeks)
Population: All subject enrolled in Step 2.
Measure: Number; unit: participants
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 16
participants | 13

4. Secondary Outcome: The Proportion of All Subjects With HCV Viral Load < 60 IU/mL at Week 72of Step 2.
Time Frame: Week 72 of Step 2
Population: All enrolled subjects.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 19
proportion of participants | 0.053 [0.001 to 1]
Statistical Analysis 1: Comparison: PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2); The proportion of subjects responding was compared to a historical null rate of 0.02. The hypothesized response rate was 0.15; Test type: Superiority or Other; p = 0.42, Exact test of proportions — This is an unadjusted p-value. Statistical significance was defined a priori as 0.10; proportion = 0.053, 90% CI 1-sided [lower limit 0.001]

5. Secondary Outcome: Absolute Change From Entry to Week 24 of Step 1 in AST and ALT.
Time Frame: From Entry to Week 24 of Step 1
Population: Subjects with both Entry and Week 24 LFT results.
Measure: Median (Inter-Quartile Range); unit: x ULN
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 17
x ULN
  24 week change in ALT (n=17) | -0.14 [-0.47 to 0.02]
  24 week change in AST (n=17) | -0.20 [-0.29 to -0.08]

6. Secondary Outcome: Absolute Change From Entry to Week 24 of Step 1 in Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR)
Time Frame: From Entry to Week 24 of Step 1
Population: Subjects with both Entry and Week 24 HOMA-IR results.
Measure: Median (Inter-Quartile Range); unit: mg/dL x uIU/mL / 405
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 16
mg/dL x uIU/mL / 405 | -1.2 [-3.6 to 0.9]

7. Secondary Outcome: Absolute Change From Entry to Week 24 of Step 1 in Fasting Total Cholesterol and Triglycerides.
Time Frame: From Entry to Week 24 of Step 1
Population: Subjects with both Entry and Week 24 fasting lipid results.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Number analyzed (Participants) | 16
mg/dL
  24 week change in total cholesterol (n=16) | 5.5 [-2.0 to 20.5]
  24 week change in triglycerides (n=16) | 28.5 [-15.5 to 73.0]

ADVERSE EVENTS:
Arm/Group | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2)
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2) (N=19)
Pancreatitis (Gastrointestinal disorders) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PIO (Step 1) Then PIO+PEG-INF+RBV (Step 2) (N=19)
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Eye pain (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Leukoplakia oral (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 6
Irritability (General disorders) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Bartholin's abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Oesophageal candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 16
Blood albumin abnormal (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 3
Blood bicarbonate abnormal (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood glucose abnormal (Investigations) | 11
Blood glucose decreased (Investigations) | 1
Blood glucose increased (Investigations) | 3
Blood phosphorus decreased (Investigations) | 2
Blood sodium decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 7
Lipase abnormal (Investigations) | 1
Lipase increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 12
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cervicobrachial syndrome (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Anger (Psychiatric disorders) | 1
Anhedonia (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Depressive symptom (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Vulvovaginal swelling (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study did not fully enroll and the small sample size precluded subgroup analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No